CLINICAL TRIAL: NCT03644524
Title: Heat Therapy and Cardiometabolic Health in Obese Women
Acronym: CMH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Christopher T Minson, PhD, Kenneth & Kenda Singer Endowed Professor, University of Oregon
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 08282015.026
Record Dates: First submitted 2018-08-20; First posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Obesity; Polycystic Ovary Syndrome; Prehypertension; PreDiabetes; Cardiovascular Risk Factor; Metabolic Syndrome
Keywords: heat therapy; blood pressure; oral glucose tolerance test; adipose tissue; muscle sympathetic nerve activity
MeSH Terms: conditions — Obesity; Polycystic Ovary Syndrome; Prehypertension; Prediabetic State; Metabolic Syndrome; Hyperthermia | interventions — Diathermy

STUDY DESIGN:
Intervention Model Description: Subjects were matched for age and BMI, then assigned to either a heat therapy intervention or time control (no intervention, just outcomes assessment at matched timepoints).
Who Masked: Outcomes Assessor
Masking Description: It was not possible to blind the subject or PI to treatment group, but all measures that were collected were analyzed offline by a blinded investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heat Therapy (Experimental): Subjects assigned to heat therapy underwent 30 1-hour hot tub sessions over 8-10 weeks (3-4 per week). The hot tub was set to 40.5 Celsius, and core temperature and heart rate were monitored throughout each session.Subjects were instructed to not make any other dietary or lifestyle changes.Cardiovascular and metabolic health assessments were made Pre (0 heat sessions), mid (after 14-16 heat sessions, ~4-5 weeks), and post (after all 30 heat sessions; ~8-10 weeks).
  Interventions: Behavioral: Heat therapy
- Time Control (No Intervention): Subjects were monitored at matched timepoints (start of study, 4-5 weeks, and 8-10 weeks) but not exposed to any intervention. Subjects were instructed to not make any dietary or lifestyle changes.

INTERVENTIONS:
Behavioral: Heat therapy — Regular hot tub use
  Arms: Heat Therapy

SUMMARY:
Traditional medical treatments are often based on research done exclusively in males, and recent research efforts in the physiology community have highlighted critical sex differences in disease presentation and progression. For example, the relative risk of fatal heart disease is 50% greater in obese, diabetic women as compared to their male counterparts, and women appear to respond differently to lifestyle interventions such as exercise compared with men. Chronic passive heat exposure (hot tub use) provides alternative or supplemental therapeutic potential for improving cardiovascular and metabolic health in obese women. In addition, passive heat exposure may offer specific cellular protection from stresses like a lack of blood flow (ischemia), which is the primary cause of fatal coronary heart disease. This study is investigating the possible cardiovascular and metabolic health benefits of chronic passive heat exposure, and whether regular hot tub use (3-4 days per week for 8-10 weeks) may reduce obese womens' cardiometabolic risk. The investigators are examining cardiovascular health through blood pressure, blood vessel stiffness, sympathetic ('fight or flight') activity, and responsiveness to stresses like increased or decreased blood flow. The investigators are also examining metabolic health through an oral glucose tolerance test and a subcutaneous fat biopsy. The goal of this research is to develop a therapy targeted toward the specific health needs and complications of obese women, in an effort to improve cardiovascular and metabolic health and provide therapeutic alternatives in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40
* Body mass index (BMI) between 30-45 kg/m2.
* Willing to maintain consistent diet and activity patterns through the study
* Willing to refrain from food, physical activity, supplements, and medications as required before testing days
* Willing to refrain from blood donations over the course of the study

Exclusion Criteria:

* overt cardiovascular disease or diabetes
* medications that affect blood vessel function (i.e. Spironolactone), insulin sensitivity (Metformin), or blood coagulation (i.e. Warfarin)
* Recent rectal, anal, or vaginal surgery
* pregnant, breastfeeding, or trying to conceive within 6 months.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
systolic blood pressure | through study completion, an average of 10 weeks
  Resting supine blood pressure, measured in triplicate with median recorded
diastolic blood pressure | through study completion, an average of 10 weeks
  Resting supine blood pressure, measured in triplicate with median recorded
oral glucose tolerance test | through study completion, an average of 10 weeks
  glucose and insulin responses to a 75-g, 2-hr oral glucose tolerance test after a 12+hr fast

SECONDARY OUTCOMES:
muscle sympathetic nerve activity burst frequency | through study completion, an average of 10 weeks
  recording of sympathetic nerve traffic during supine rest, quantified as burst count per minute
arterial wall thickness (carotid) | through study completion, an average of 10 weeks
  intimal thickness of common carotid artery assessed using doppler ultrasonography
arterial wall thickness (femoral) | through study completion, an average of 10 weeks
  intimal thickness of superficial femoral artery assessed using doppler ultrasonography
dynamic arterial compliance (carotid) | through study completion, an average of 10 weeks
  arterial compliance of common carotid artery measured using ultrasonography
dynamic arterial compliance (femoral) | through study completion, an average of 10 weeks
  arterial compliance of superficial femoral artery measured using ultrasonography
flow mediated dilation | through study completion, an average of 10 weeks
  flow-mediated dilation of brachial artery, expressed as % change in diameter. A measure of endothelial function.
flow mediated dilation after ischemia-reperfusion | through study completion, an average of 10 weeks
  flow-mediated dilation of brachial artery, expressed as % change in diameter, following 20 minute ischemia-20 minute reperfusion. A measure of vascular tolerance to ischemia-reperfusion stress.
Abdominal subcutaneous fat biopsy | through study completion, an average of 10 weeks
  Adipose tissue sample analyzed for insulin signaling, markers of inflammation, and heat shock protein expression

OTHER OUTCOMES:
C-reactive protein | through study completion, an average of 10 weeks
  serum measurement of high-sensitivity C-reactive protein, global inflammatory marker
Cholesterol panel | through study completion, an average of 10 weeks
  serum measurement of cholesterol

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No